CLINICAL TRIAL: NCT00653510
Title: The Effect of Acute Hyperglycemia on Cardiac Output, Amino Acid, Lipid and Glucose Metabolism in Patients With Type 2 Diabetes
Brief Title: The Metabolic Effects of Acute Hyperglycemia in Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Regionshospitalet Silkeborg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: UK-M20070267
Record Dates: First submitted 2008-03-25; First posted 2008-04-07 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2012-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes; Dysregulation; Metabolism; Cardiac output
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Euglycemic (Experimental): The patients will be examined with a blood glucose at around 5-7 mmol/L.
  Interventions: Drug: Actrapid (human insulin)
- Hyperglycemic (Experimental): The patients will be examined with a blood glucose at around 18-20 mmol/L
  Interventions: Drug: Actrapid (human insulin)

INTERVENTIONS:
Drug: Actrapid (human insulin) — On day one the patients will receive glucose and insulin in order to reach a blood sugar around 18 and 20 mmol/L and on day two the patients will receive glucose and insulin in order to have a blood sugar around 5 and 7 mmol/L. On both days amino acid, lipid and glucose metabolism will be assessed by means of whole body isotope dilution.

SUMMARY:
The purpose of the study is to characterize the changes in amino acid, lipid and glucose metabolism in patients with type 2 diabetes exposed to acute hyperglycemia. Moreover we wish to assess the effect of acute hyperglycemia on cardiac output.

DETAILED DESCRIPTION:
Cardiovascular disease is the main cause of death in modern Western societies. Obesity, diabetes and the metabolic syndrome are the main risk factors for cardiovascular disease. People with type 2 diabetes and no history of heart disease have a risk of myocardial infarction similar to the risk in non-diabetic patients with known heart disease.

However, the causal relationship between obesity, diabetes and cardiovascular disease is unclear. Insulin resistance leads to many metabolic abnormalities, including high circulating levels of free fatty acids (FFA). FFA induces insulin resistance and may lead to beta cell failure. In addition FFA may directly worsen the metabolic and electrochemical performance of the working heart. Moreover it is still unclear how acute hyperglycemia affects cardiac output.

In this study our purpose is to characterize the changes in amino acid, lipid and glucose metabolism in patients with type 2 diabetes exposed to acute hyperglycemia (blood glucose between 18 and 20 mmol/L) compared to the amino acid, lipid and glucose metabolism at a normal glucose level (blood glucose between 5 and 7 mmol/L). The results from the patients with type 2 diabetes will be compared with results from healthy controls examined in a fasting basal state. The patients must not suffer from any kind of serious heart disease and should be treated with insulin.

Moreover we wish to compare cardiac output at high and normal blood glucose levels, respectively. Cardiac output will primarily be assessed by doppler echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Written consent
* Age 40-75 years old
* BMI between 22 and 35
* Type 2 diabetes treated with insulin (< 60 IE/day)

Exclusion Criteria:

* Severe disease
* Severe cardiac disease

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-03; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Metabolic changes | 6 hours

SECONDARY OUTCOMES:
Left ventricular function | 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Niels Moeller, Professor, Principal Investigator — Department M (Endocrinology and diabetes), Aarhus University Hospital, Nørrebrogade 44, 8000 Århus C, Denmark
Locations (1):
- Department M (Endocrinology and Diabetes), Aarhus University Hospital, Aarhus, Aarhus, Denmark

REFERENCES:
- [Derived] Nielsen R, Norrelund H, Kampmann U, Botker HE, Moller N, Wiggers H. Effect of acute hyperglycemia on left ventricular contractile function in diabetic patients with and without heart failure: two randomized cross-over studies. PLoS One. 2013;8(1):e53247. doi: 10.1371/journal.pone.0053247. Epub 2013 Jan 8. PMID 23308171
- [Derived] Nielsen TS, Kampmann U, Nielsen RR, Jessen N, Orskov L, Pedersen SB, Jorgensen JO, Lund S, Moller N. Reduced mRNA and protein expression of perilipin A and G0/G1 switch gene 2 (G0S2) in human adipose tissue in poorly controlled type 2 diabetes. J Clin Endocrinol Metab. 2012 Jul;97(7):E1348-52. doi: 10.1210/jc.2012-1159. Epub 2012 Apr 24. PMID 22535977